CLINICAL TRIAL: NCT02003378
Title: Comparison of Physiologic Response With Rate Adaptive Pacing Driven by Minute Ventilation and Accelerometer
Acronym: RAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albany Medical College (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Sujata S. Balulad, MD, Principal Investigator, Albany Medical College
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RAP
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Chronotropic Incompetence
Keywords: Chronotropic incompetence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minute Ventilation (MV) (Active Comparator): Pacemaker sensor set to MV (Cross over study)
  Interventions: Device: Pacemaker sensor set to MV
- Accelerometer (XL) (Active Comparator): Pacemaker sensor set to XL (Cross over study)
  Interventions: Device: Pacemaker sensor set to XL

INTERVENTIONS:
Device: Pacemaker sensor set to MV — Pacemaker sensor set to minute ventilation
  Arms: Minute Ventilation (MV)
Device: Pacemaker sensor set to XL — Pacemaker sensor set to accelerometer
  Arms: Accelerometer (XL)

SUMMARY:
Some patients' heart rates do not increase as needed during activities and exercise, which can make them feel tired and fatigued easily. The patients in this study have a pacemaker with a FDA approved rate response sensor, which senses activity level by sensing motion (through a component known as an accelerometer) and/or breathing changes (known as minute ventilation). These changes in motion or breathing make the pacemaker increase the patient's heart rate. This study is being conducted to see which rate response sensor is better (motion driven or breathing driven). The study is also investigating whether optimizing the sensor based on the individual patient will give better results in terms of increasing the patient's exercise capacity. The hypothesis is that rate responsive pacing driven by the minute ventilation sensor results in improved functional capacity compared to accelerometer in chronotropically incompetent patients.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, two-arm (with crossover to other arm) trial that will investigate the benefit of rate responsive pacing with either MV or XL in pacemaker patients that have chronotropic incompetence (CI). Blinding will occur for both the patient and the research personnel who are collecting primary endpoint data. The study will enroll patients that have an implanted dual/single chamber pacemaker, which has both the minute ventilation (MV) and accelerometer (XL) rate-adaptive sensors.

The initial study visit called as baseline visit for newly implanted patients (at 2 weeks from implant) and for previously implanted patients (at the time of enrolling in the study).

Patients will complete a 6-min walk test at the baseline study visit to screen for CI based on the intrinsic heart rate achieved during the walk while pacemaker set to DDD/VVI with both sensors set to passive. All patients that are enrolled in the study will get treadmill exercise stress test by chronotropic assessment exercise protocol (CAEP) to confirm CI. Patients will be determined to have CI by completing a maximal effort exercise treadmill stress test with peak perceived exertion by Borg scale of >16 (18) with the pacemaker programmed to DDD/VVI with both device sensors set to passive. Patients that do not meet the criteria of CI after CAEP treadmill test will not continue in the trial.

Patients that have CI will then be randomized in a 1:1 ratio to programming the rate-adaptive sensor to either MV or XL. The MV or XL rate-adaptive sensor will be optimized for each patient using stress test derived age predicted maximum heart rate by adjusting response factor to achieve MCR slope of 1.

At the 4-week visit, patients that have CI will complete a second CAEP treadmill test in their randomized setting with pacer set as DDDR/VVIR. They will also complete 6-minute walk test and pacemaker interrogation. They will be crossed over to the other sensor group at this time by changing the sensor setting.

At 8 week visit, patients will have another CAEP treadmill test, 6-minute walk test and pacemaker interrogation in their randomized crossed over group setting.

Patients that have CI will get quality of life assessment using SF-36 questionnaire and Aquarel questionnaire at baseline visit, 4 and 8 week visit in their randomized setting.

ELIGIBILITY:
Inclusion Criteria:

* Willing and capable of providing informed consent for participation
* Previously received, or previously scheduled to receive, dual-chamber/single chamber pacemaker with active atrial and ventricular leads.Boston Scientific Ingenio K172, K173, K174; or (both Ingenio and Advantio have similar rate response features) Advantio K062, K063, K064 (Boston Scientific CRM, St. Paul, MN).
* Plans to remain in the long-term care of his/her enrolling physician and is available for study follow-up for three months post-enrollment
* Patients with or without one or more of the following are permitted to enroll:
* Sinus node dysfunction with pacemaker
* Mobitz II second degree heart block or third degree heart block with pacemaker
* Chronic atrial fibrillation and other atrial arrhythmias with controlled heart rate within the past 90 days prior to consent
* Paroxysmal atrial fibrillation on rate controlling medication as long as same rhythm stays throughout the study, sinus or atrial fibrillation.
* Patients with pacemakers requiring beta blocker (or other rate limiting medications) therapy

Exclusion Criteria:

* Neuromuscular, orthopedic, or vascular disability that prevents normal walking (e.g., intermittent claudication, arthritis, residual stroke weakness, need for a wheelchair or walker)
* A symptom-limited exercise protocol is thought to be dangerous or contra-indicated, including but not limited to changing pattern of chest discomfort, unstable angina or uncontrolled arrhythmias Severe pulmonary disease with inability to exercise
* Severe heart failure with dyspnea at rest and inability to exercise (NYHA class IV) and qualify for the CRT-D
* Life expectancy is less than 12 months due to other medical conditions, per physician discretion
* Has or indicated for an implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy-defibrillator (CRT-D)
* Currently, or within 30 days prior to consent, enrolled in another investigational study that would directly impact the treatment or outcome of the current study.
* Younger than 18 years of age
* Patients with pacemakers of unipolar atrial or ventricular lead configuration
* Patients with abdominal pacemaker implants
* Patients on a ventilator
* Patients with a pacemaker with epicardial lead
* Patients with Pneumothorax, pericardial effusion or pleural effusion
* Pregnant or planning to become pregnant during the study (method of assessment upon physician's discretion). Pregnancy test will be done for all female patients of childbearing age before the study, and at each visit.
* Unable or unwilling to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Metabolic chronotropic relationship (MCR) slope | 2 weeks, 6 weeks, and 10 weeks post-implant/post enrollment
  Improvement in functional capacity, determined by MCR slope - if greater using the minute ventilation senor of the accelerometer sensor in patients with chronotropic incompetence

SECONDARY OUTCOMES:
Changes in heart rate and distance covered during 6-minute walk test | 2 weeks, 6 and 10 weeks post-implant/post enrollment
  To evaluate the superiority of the minute ventilation sensor or the accelerometer sensor by comparing changes in heart rate and distance covered during activities using a 6 minute walk test.
Exercise time during chronotropic assessment exercise protocol (CAEP) stress test | 2 weeks, 6 and 10 weeks post-implant/post enrollment
  To evaluate the superiority of the minute ventilation sensor or the accelerometer sensor related to exercise time during the CAEP stress test
Quality of life (QOL) assessment | 2 weeks, 6 and 10 weeks post-implant/post enrollment
  SF-36 questionnaire and Aquarel questionnaire to assess quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Sujata Balulad, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical College, Albany, New York, United States